CLINICAL TRIAL: NCT00359333
Title: Multiple Centers, Prospective, Phase II Trial of Gemcitabine and Docetaxel Combination Chemotherapy in Patients With Locally Advanced/Metastatic Soft Tissue Sarcoma or Imatinib Mesylate Refractory Advanced/Metastatic Malignant Gastrointestinal Stromal Tumor
Brief Title: Phase II Trial of Locally Advanced/Metastatic Soft Tissue Sarcoma or Advanced/Metastatic Malignant GIST
Acronym: STS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Mackay Memorial Hospital (Other); Tri-Service General Hospital (Other); China Medical University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Taichung Veterans General Hospital (Other); Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1706
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Sarcoma; Malignant Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: Gemcitabine , Docetaxel

INTERVENTIONS:
Drug: Gemcitabine , Docetaxel — Gemcitabine 800 mg/m2 IV over 80 minutes on day 1 and day 8, and Docetaxel 60 mg/m2 IV over 60 minutes on day 1 of a 21-day cycle

SUMMARY:
Study Design Type of Study This is an open-label, single arm, prospective, multiple-center phase II study

Duration of the Study Period in One Subject Treatment duration is planned for six cycles, unless there is evidence of disease progression or unacceptable toxicity. Patients with continued response after six cycles could receive two additional cycles of therapy. In case complete response and in the absence of unacceptable toxicity, treatment will be continued for at least 2 further cycles to achieve the minimal of 6 total cycles.

Study Objectives Primary Objective The primary objective is to determine the response rate of sequential gemcitabine and docetaxel combination in patients with locally advanced/metastatic soft tissue sarcoma or imatinib mesylate refractory GIST.

Secondary Objectives The secondary objectives of this study are to determine the time to progression in patients treated with this regimen, the toxicity of this regimen in these patients, the overall survival and the quality of life.

Molecular analysis of genetic aberration in soft tissue sarcoma The genetic aberrations of soft tissue sarcoma as reported in literature will be determined. The genetic aberration will be correlated to chemotherapy responses.

c-kit and PDGFR gene mutations induced by imatinib mesylate and chemotherapy Those acquired gene mutation of c-kit and PGDFR induced by imatinib mesylate will be first determined. We will also examine further gene mutation of c-kit and PGDFR caused by combination chemotherapy.

DETAILED DESCRIPTION:
Eligibility Criteria:

Inclusion criteria:

Patients must have a histologically confirmed diagnosis of (1) locally advanced unresectable or metastatic soft tissue sarcoma; or (2) unresectable/metastatic GIST previously treated with imatinib mesylate and is documented to have drug resistance to imatinib mesylate treatment defined by tumor progression.

Age greater than or equal to 18 years and younger than or equal to 70 years old.

Measurable disease: defined as lesions that can be measured in at least one dimension by physical examination or medical imaging techniques. Ascites, pleural effusions, and bone marrow disease will not considered measurable disease.

Patients must have an ECOG performance status of less than or equal to 2. Patients must have recovered (defined as toxicity less than grade 2) from toxic effects of all prior therapy before entering onto study.

A treatment of drug free interval of at least 4 weeks since the last dose of chemotherapy or imatinib mesylate therapy is required.

More than 4 weeks since prior radiotherapy is required. Adequate bone marrow function with an ANC greater than or equal to 1,500/ml, platelet count greater than or equal to 100,000/ ml (transfusion independent) and hemoglobin greater than or equal to 8.0 g/dl (transfusions permitted).

Patients must have adequate renal function with serum creatinine less than or equal to 1.5 mg/dl.

Patients must have adequate liver function, defined as bilirubin within 1.5 times the upper limit of normal, and liver transaminases within 2.5 times the upper limit of normal.

All patients must sign a document of informed consent indicating their awareness of the investigational nature and the risks of the study.

Exclusion criteria:

Patients who have prior treatment with gemcitabine or taxane. Pregnant or breast feeding females. Active or uncontrolled infection. Patients with brain or leptomeningeal metastases.

Treatment Plan:

For safety and convenience of drug administration, a Port-A catheter implantation is required before the start of the first chemotherapy course.

Gemcitabine 800 mg/m2 will be administered by intravenous infusion over 80 minutes on day 1 and day8, and docetaxel 60 mg/m2 over 60 minutes on day 1 of a 21-day cycle. After the first cycle of the chemotherapy, if the ANC of the patient is always ≥ 1500/ml before the starting of the next cycle, the dosage of docetaxel will be escalated to 75 mg/m2 on day 1 of the next and following cycles.

All patients received filgrastim 300 mg subcutaneously once per day on day 12 to 15.

During treatment, complete blood cell counts are performed weekly. History and physical examinations and assessment of toxicities are performed before each cycle of treatment.

Patients with progressive disease evaluated at the third or sixth course should be suggested salvage treatment and withdrawn from protocol treatment.

Patients with SD, CR, or PR continue on study and undergo repeat CT scan after cycle 6.

Patients who have continued response at the sixth course will be given two additional courses of chemotherapy, and undergo a CT scan again after cycle 8.

Dose Adjustments: dose adjustments were required in the following situations:

If patients experienced febrile neutropenia or had platelet count of less than 25,000/ml lasting more than 5 days, doses of gemcitabine and docetaxel will be reduced to 75% of the previous dose in all subsequent cycles.

If at day 1 of the treatment cycle the ANC is less than 1,500/ml or if the platelet count is less than 50,000/ml, treatment will be delayed 1 week.

Patients in whom the ANC or platelet count has not recovered after a 2-week delay will be removed from the study.

If on day 8 the ANC is 500 to 999/ul and the platelet is ≥ 50,000/ul, gemcitabine are provided at 75% of the day 1 doses.

If at day 8 the ANC is less than 500/ul or if the platelet count is less than 50,000/ul, gemcitabine at the day 8 dose will not be provided in that cycle.

If the patients experience grade 3 or 4 neurotoxicity, treatment will be delayed for 1 week. If neurotoxicity has resolved to ≤ grade 2, treatment resumed with the docetaxel dose decreases to 75% of the previous dose for all subsequent cycles.

If the patient's bilirubin level is more than 1.5 mg/dL, the docetaxel treatment will be hold for that cycle. If bilirubin returns to ≤ 1.5 mg/dL, docetaxel treatment will be resumed in the subsequent cycles.

If patients experienced other grade 3 or 4 nonhematologic toxicities (except alopecia), treatment will be hold for up to 2 weeks; treatment will be resumed if nonhematologic toxicity has resolved to ≤ grade 2.

Criteria for Withdrawal from Study Documented disease progression. A new cycle of chemotherapy will be given if ANC ≥ 1500/ml, platelet count ≥ 50,000/ ml (transfusion independent) and hemoglobin ≥ 8.0 g/dl (transfusions permitted). On the scheduled Day 1 of a new treatment cycle, if the hemogram is not yet recovered, chemotherapy will be postponed and the patient will be followed weekly until the resolution of toxicity. If the interruption is more than 2 weeks from the schedule Day 1, the patient should be taken off protocol treatment.

Occurrence of adverse event that the attending physician considers withdrawal from protocol treatment is for the patient's optimal benefit.

Voluntary withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* 5.1.1 Patients must have a histologically confirmed diagnosis of (1) locally advanced unresectable or metastatic soft tissue sarcoma; or (2) unresectable/metastatic GIST previously treated with imatinib mesylate and is documented to have drug resistance to imatinib mesylate treatment defined by tumor progression.

5.1.2 Age greater than or equal to 18 years and younger than or equal to 70 years old.

5.1.3 Measurable disease: defined as lesions that can be measured in at least one dimension by physical examination or medical imaging techniques. Ascites, pleural effusions, and bone marrow disease will not considered measurable disease.

5.1.4 Patients must have an ECOG performance status of less than or equal to 2. 5.1.5 Patients must have recovered (defined as toxicity less than grade 2) from toxic effects of all prior therapy before entering onto study.

5.1.6 A treatment of drug free interval of at least 4 weeks since the last dose of chemotherapy or imatinib mesylate therapy is required.

5.1.7 More than 4 weeks since prior radiotherapy is required. 5.1.8 Adequate bone marrow function with an ANC greater than or equal to 1,500/ml, platelet count greater than or equal to 100,000/ ml (transfusion independent) and hemoglobin greater than or equal to 8.0 g/dl (transfusions permitted).

5.1.9 Patients must have adequate renal function with serum creatinine less than or equal to 1.5 mg/dl.

5.1.10 Patients must have adequate liver function, defined as bilirubin within 1.5 times the upper limit of normal, and liver transaminases within 2.5 times the upper limit of normal.

5.1.11 All patients must sign a document of informed consent indicating their awareness of the investigational nature and the risks of the study.

Exclusion Criteria:

* 5.2.1 Patients who have prior treatment with gemcitabine or taxane. 5.2.2 Pregnant or breast feeding females. 5.2.3 Active or uncontrolled infection. 5.2.4 Patients with brain or leptomeningeal metastases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Tumor response | CT scan are repeated after every 3 courses of chemotherapy. Patients who complete at least two courses of chemotherapy are eligible for evaluating response.

SECONDARY OUTCOMES:
Time to tumor progression Overall survival Quality of life | Evaluable for toxicity if they received at least one dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jer Huang, Principal Investigator — Mackay Memorial Hospital; Li-Tzong Chen, PHD, Principal Investigator — National Health Research Institutes, Taiwan; Chung- Huang Chan, PHD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan